CLINICAL TRIAL: NCT00662454
Title: Oral Contraceptive Efficacy and Body Weight: Does Obesity Affect the Risk of Contraceptive Failure?
Brief Title: Oral Contraceptive Efficacy and Body Weight
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Oregon Health and Science University (Other)
Collaborators: National Institutes of Health (NIH) (NIH); Oregon Clinical and Translational Research Institute (Other)
Responsible Party: Principal Investigator, Alison Edelman, Principal Investigator, Oregon Health and Science University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: OHSU FAMPLAN 0411; NIH R03 HD053611 01
Record Dates: First submitted 2008-04-16; First posted 2008-04-21 (Estimated); Last update posted 2020-09-16 (Actual); Status verified 2020-09

CONDITIONS: Contraception; Body Weight
Keywords: contraceptive; efficacy; body weight
MeSH Terms: conditions — Body Weight | interventions — Ethinyl Estradiol-Norgestrel Combination

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- I (Active Comparator): 10 normal weight women (BMI < 25 kg/m2)
  Interventions: Drug: ethinyl estradiol / levonorgestrel
- II (Active Comparator): 10 obese women (BMI >30 kg/m2)
  Interventions: Drug: ethinyl estradiol / levonorgestrel

INTERVENTIONS:
Drug: ethinyl estradiol / levonorgestrel — Take one tablet daily of 20 mcg ethinyl estradiol/100 mcg levonorgestrel for 21 days plus 7 days of placebo tablets, repeat for two months total duration.
  Other Names: Alesse
  Arms: I
Drug: ethinyl estradiol / levonorgestrel — Take one tablet daily of 20 mcg ethinyl estradiol/100 mcg levonorgestrel for 21 days plus 7 days of placebo tablets, repeat for two months total duration.
  Other Names: Alesse
  Arms: II

SUMMARY:
The purpose of the blood spot validation portion of the study is to test if measuring female hormone levels in the blood is as accurate through a finger stick, as it is by a blood draw from a vein. The purpose of the feasibility study is to evaluate ovulation occurrence in two populations of oral contraceptive users: heavier and lighter women.

DETAILED DESCRIPTION:
The blood spot validation portion of the study tests the hypothesis that progesterone assays from self-collected daily blood spots are equivalent to serum samples, and that the values obtained can identify women that ovulate. After validating collection methods, enrollment will begin for the feasibility portion of the study looking at thin and heavy women on birth control pills. All women in this portion of the study will take a very-low dose birth control pill that is normally available through a doctor's office. During each month of the study, women will have their blood pressure and weight recorded, and have their blood drawn twice per week or use a finger stick kit daily at home to check for the natural hormones and brain chemicals that tells if an egg develops. During the last week of each menstrual cycle (period week), women will also have their blood drawn to measure the levels of hormone found in the birth control pill. Women will also need to report in a written diary that they have taken their birth control pill for the day.

ELIGIBILITY:
Inclusion Criteria:

* age 18 to 35
* single baseline hematocrit ≥ 36%
* single progesterone level of 3 ng/mL or greater during the luteal phase (days 18 to 25) in the menstrual cycle prior to treatment with OCs.

Exclusion Criteria:

* any absolute contraindications to ethinyl estradiol and levonorgestrel
* smoking
* actively seeking or involved in a weight loss program (must be weight stable)
* pregnancy, breastfeeding, or seeking pregnancy
* diagnosis of Polycystic Ovarian Syndrome
* recent (8 week) use of OC (patch or ring included), intrauterine, or implantable hormonal contraception
* DepoProvera use within six months
* current use of drugs that interfere with metabolism of sex steroids.

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 120 (Actual)
Dates: Start 2006-01; Primary Completion 2006-05 (Actual); Study Completion 2006-05 (Actual)

PRIMARY OUTCOMES:
Concentrations of circulating oral contraceptives dosed in a standard cyclic fashion in obese and normal BMI cohorts | Approximately one year

CONTACTS AND LOCATIONS:
Overall Officials: Alison Edelman, MD, MPH, Principal Investigator — Oregon Health and Science University
Locations (1):
- Oregon Health & Science University, Portland, Oregon, United States

REFERENCES:
- See also: OHSU Women's Health Research Unit — http://www.ohsuwomenshealth.com/research/index.html